CLINICAL TRIAL: NCT02533622
Title: A Clinical Study Of The Impact Of Total Care® Bed System Combined With The Liko Lift to Facilitate Early Progressive Mobility Compliance and Associated Clinical and Financial Outcomes.
Brief Title: Holy Name Progressive Mobility in the ICU
Status: Completed | Type: Observational
Sponsor: Hill-Rom (Industry)
Responsible Party: Sponsor
Other Study IDs: QI-2010-05
Record Dates: First submitted 2012-03-22; First posted 2015-08-27 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Respiratory Failure
Keywords: progressive mobility
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard of care: Patients admitted to the ICU will receive current standard of care related to mobility
- Progressive mobility: patients admitted to the ICU will receive mobility per Progressive Mobility protocol using TotalCare beds and lifts

SUMMARY:
Despite the known complications of immobility for ICU patients, compliance to mobility protocols is lacking in many institutions. Significant barriers have been described to compliance to up in chair and weight bearing orders in the ICU. Recent studies indicate that if progressive mobility is performed for acutely ill ICU patients they may have a reduced ICU length of stay, reduced overall hospital length of stay, incur lower hospital costs, and reduce the rate of some medical complications and increase functionality post ICU discharge.

The current protocol seeks to understand whether or not the TotalCare® P500 Bed System and the Liko Lift can remove some of the barriers associated with progressive mobility compliance.

DETAILED DESCRIPTION:
This study is designed as a process improvement program to increase compliance to a progressive mobility protocol in an ICU setting. The first part of the study (4-6 months period depending on time required for implementation) will document 1st day of weight bearing as well as the secondary outcome measures of this of progressive mobility protocol as are currently in place in the ICU for patients that meet the inclusion/exclusion criteria. Ease of progressive mobility implementation will be assessed. Appropriate education will be performed as to the importance of progressive mobility.

The second part of the study (4-6 months) will document the same outcomes, however, the progressive mobility protocol will now include a standardized process using the Total Care® P500 Bed System combined with the Liko Lift. During the second study period, patients will progress in a stepped protocol (see section 6.2) beginning with head of bed (HOB) at 30o to initiate orthostatic stress three times daily with increasing time intervals, then increasing HOB angle, time, and finally to standing and bearing weight. The Total Care® P500 Bed System and the Liko Lift will be placed on all participating units for the duration of the second phase of the study.

Compliance to specific outcome measures again will be measured as well as the ease of Progressive Mobility implementation. The total study period will be 8-12 months (allowing time for bed delivery and education).

Patients who meet the inclusion/exclusion criteria for study will be enrolled. Protocol based "up in chair" and "standing" orders will be followed for compliance, and length of actual sitting in full chair or standing. If patients undergo "full chair" in the bed, this will be considered "up in chair." Time/days to first weight bearing, as defined as weight bearing in a standing position for at least 1 minute will be documented. ICU LOS, Ventilator Days will be assessed at ICU discharge for study patients. Nursing satisfaction and ease of PM protocol adherence surveys will be performed after each study period and will assess both standard of care and Total Care® bed/Liko lift systems.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years old.
* Patient has been admitted to the ICU for less than 3 days prior to study enrollment
* Patients require mechanical ventilation for > 48 hours

Exclusion Criteria:

* Patient has an unstable spinal injury.
* Patient weighs less than 70 pounds or more than 450 pounds
* Mobilization is contraindicated by Patient's condition. Such as hip fractures or other injury that would impede standing posture.
* Patient was unable to walk without assistance prior to ICU admission.
* Patient was cognitively impaired prior to ICU admission.
* Patient has experienced acute stroke with neurologic impairment
* Patient's primary diagnosis is drug overdose.
* Patient has Comfort Care Measures/End of Life orders and/or is at an end stage terminal disease state.
* Patient requires a bed other than the standard care bed for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the Medical ICU
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
First out of bed, which is to be defined as the first time that a patient stands whether assisted or not for > 1 minute. | at ICU discharge (current avg LOS = 6 days)

SECONDARY OUTCOMES:
ICU length of stay | at ICU discharge (current avg LOS = 6 days)
Days of Mechanical Ventilation assessed as time to extubation. Extubation is to be defined as the time when the ET tube is removed from the airway | at ICU discharge (current avg LOS = 6 days)
Compliance with, Number and Duration of Up in Chair episodes. Patients will be considered compliant if they complete 100% of prescribed episodes. | at ICU discharge (current avg LOS = 6 days)
ICU readmission rate (within 30 days) | at ICU discharge (current avg LOS = 6 days)
Incidence of nosocomial pressure ulcers and change in existing pressure ulcers | at ICU discharge (current avg LOS = 6 days)
Nursing satisfaction and ease of use for each bed system for the purpose of mobilizing patients | at ICU discharge (current avg LOS = 6 days)
Financial outcomes will be calculated if any reduction in days / hours of mechanical ventilation and days of ICU admission occur | at ICU discharge (current avg LOS = 6 days)

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Tracy, RN, MSN, Principal Investigator — Holy Name Hospital
Locations (1):
- Holy Name Medical Center, Teaneck, New Jersey, United States